CLINICAL TRIAL: NCT02368015
Title: An Explorative Study Determining the Hepatic Cyst Penetration of Cefazolin and Factors Affecting Penetration.
Brief Title: Penetration of Cefazolin Into Hepatic Cysts
Acronym: PENTAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NL49426.091.14
Record Dates: First submitted 2014-12-29; First posted 2015-02-20 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Hepatic Cyst
Keywords: Penetration; Cefazolin; Hepatic cyst
MeSH Terms: interventions — Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with a large hepatic cyst (Other): During this study all subjects undergo aspiration sclerotherapy and receive antibiotic prophylaxis with a single dose of cefazolin (intravenous infusion 1000mg) following standard care.
  In order to secure patient safety and allow accurate measurement of cefazolin concentrations, an additional peripheral intravenous cannula (IVC) will be placed to allow blood withdrawal at three timepoints.
  Interventions: Other: Peripheral intravenous cannula (IVC); Drug: cefazolin

INTERVENTIONS:
Other: Peripheral intravenous cannula (IVC) — Blood samples will be withdrawn prior, during and after the procedure using an additional peripheral intravenous cannula (IVC).
Drug: cefazolin

SUMMARY:
Hepatic cysts are fluid-filled cavities located in the liver parenchyma. They are usually asymptomatic, but can cause mass-related symptoms as abdominal pain, dyspnea and nausea. Aspiration sclerotherapy is indicated in patients with a dominant hepatic cyst to alleviate symptoms by draining the hepatic cyst to reduce cyst diameter. Spontaneous cyst infection, or following aspiration sclerotherapy, presents a severe complication of hepatic cystic disease requiring frequent hospitalization, long-term antibiotic treatment, and in some invasive therapies. Evidence that antibiotics are able to reach adequate intracystic concentration is however lacking. To prevent procedure-related cyst infection in patients receiving aspiration sclerotherapy, cefazolin prophylaxis is given as standard of care. In this study we want to assess the hepatic cyst penetration capacity of cefazolin by comparing serum and cyst fluid concentrations of cefazolin. We hypothesize that cefazolin is able to penetrate hepatic cysts, with treatment naïve cyst allowing a better penetration, reducing the risk of developing cyst infection following aspiration sclerotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Indication for aspiration and sclerotherapy
* Providing informed consent

Exclusion Criteria:

* Presence of an arteriovenous fistula, history of mastectomy or lymph node dissection at both extremities
* Signs of phlebitis, defined as localized skin redness and swelling, at both extremities
* History of cephalosporin and/or penicillin allergy consisting of IgE-mediated reactions as anaphylaxis, angioedema, urticaria.
* Any current or prior medical condition that may interfere with the conduct of the study or the evaluation of its results in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Hepatic cyst penetration of cefazolin defined as the ratio (%) of cyst aspirate concentration (µg/ml) to serum concentration (µg/ml) of cefazolin. | Intraoperative

SECONDARY OUTCOMES:
Segmental location (I-VIII) of hepatic cyst | Baseline
Volume (mL) of hepatic cyst | Baseline
Blood parameter: total protein (g/l) | Intraoperative
Blood parameter: albumin (g/l) | Intraoperative
Blood parameter: urea (mmol/l) | Intraoperative
Blood parameter: white blood cell count (*10^9/l) | Intraoperative
Blood parameter: white blood differentiation (%) | Intraoperative
Blood parameter: CRP (mg/l) | Intraoperative
Blood parameter: direct bilirubin (µmol/L) | Intraoperative
Blood parameter: total bilirubin (µmol/L) | Intraoperative
Blood parameter: CA 19.9 (E/ml) | Intraoperative
Blood parameter: creatinine (µmol/L) | Intraoperative
Cyst fluid parameter: total protein (g/l) | Intraoperative
Cyst fluid parameter: albumin (g/l) | Intraoperative
Cyst fluid parameter: urea (mmol/l) | Intraoperative
Cyst fluid parameter: white blood cell count (*10^9/l) | Intraoperative
Cyst fluid parameter: white blood cell differentiation (%) | Intraoperative
Cyst fluid parameter: CRP (mg/l) | Intraoperative
Cyst fluid parameter: direct bilirubin (µmol/L) | Intraoperative
Cyst fluid parameter: total bilirubin (µmol/L) | Intraoperative
Cyst fluid parameter: CA 19.9 (E/ml) | Intraoperative
Cyst fluid parameter: sodium (mmol/l) | Intraoperative
Cyst fluid parameter: pH | Intraoperative
Number of patients that develop clinical signs indicating aspiration sclerotherapy-induced cyst infection | Until four weeks after aspiration sclerotherapy
Number of participants with adverse events | until four weeks after aspiration sclerotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Center; Department of Gastroenterology & Hepatology, Nijmegen, Gelderland, Netherlands